CLINICAL TRIAL: NCT06379815
Title: Effect of Oral Lactate Ingestion on Appetite Regulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Tom Hazell, Principle Investigator, Wilfrid Laurier University
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EMRL-23-03
Record Dates: First submitted 2024-04-12; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Appetitive Behavior
Keywords: lactate; appetite regulation; acylated ghrelin; energy intake
MeSH Terms: conditions — Appetitive Behavior | interventions — Sodium Lactate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will consume a sodium lactate and sodium chloride placebo in a double-blind, crossover design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The allocation of lactate and placebo will be completed by a researcher not involved in data collection. Both the participant and the researchers collecting and analyzing the data will be blinded to the treatment allocation. This will be completed in a counter-balanced order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Lactate (Experimental): Participants will received 0.45 g/kg of sodium lactate (SO179, Spectrum Chemical MFG Group) mixed with water. This will be mixed at a ratio of 30 mL per g of lactate. Lemon juice is added to the mixture at a specific ratio to balance the pH of the solution. Crystal light will also be added to avoid any taste differences between beverages.
  Interventions: Other: Sodium Lactate
- Sodium Chloride (Placebo Comparator): Participants will receive a equimolar amount of sodium chloride (S9888, MilliporeSigma) mixed with water. The amount of water, lemon juice, and crystal light will be matched to that of the sodium lactate condition.
  Interventions: Other: Sodium Chloride

INTERVENTIONS:
Other: Sodium Lactate — See arm/group description.
  Arms: Sodium Lactate
Other: Sodium Chloride — See arm/group description.
  Arms: Sodium Chloride

SUMMARY:
The goal if this study is to determine how oral lactate ingestion affects markers of appetite regulation. Researchers will compare oral lactate ingestion to a sodium chloride placebo. Participants will consume the lactate or placebo solution and then have blood samples and assessments of appetite over the course of 90 min. Free-living energy intake will be measured for 3 days surrounding each experimental session.

DETAILED DESCRIPTION:
The purpose of this study is to explore the effects of oral lactate ingestion on appetite regulation in humans. To do this males and females will report to the laboratory for 2 experimental sessions completed in a counterbalanced, double-blinded manner. During one session a lactate solution will be ingested, in another session an equimolar sodium chloride solution will be ingested that matches the osmolarity of the lactate condition. Venous blood samples and subjective appetite perceptions will be obtained at five time points during each experimental session. Energy expenditure will be measured through accelerometers placed on the participants anterior thigh by an investigator on the morning the day before the session and worn over the experimental period (day before, day of, day after) recording their physical activity. Energy intake will be tracked using a smartphone mobile application called Keenoa over the same time period the accelerometers are worn.

ELIGIBILITY:
Inclusion Criteria:

* Deemed healthy using Canadian Society for Exercise Physiology Get Active Questionnaire
* Female participants must be eumenorrheic (menstrual cycle length between 21-35 days)

Exclusion Criteria:

* Failure to meet inclusion criteria
* Taking supplements or medications known to affect metabolism (e.g., creatine, beta-blockers)
* Currently pregnant or a pregnancy of >3 months within the last 3 years,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Blood Lactate | Pre-ingestion, 30 minutes following ingestion, 45 minutes following ingestion, 60 minutes following ingestion, and 90minutes following ingestion.
  Lactate measured in blood.
Acylated ghrelin | Pre-ingestion, 30 minutes following ingestion, 45 minutes following ingestion, 60 minutes following ingestion, and 90minutes following ingestion.
  Acylated ghrelin measured in blood via ELISA.
Total ghrelin | Pre-ingestion, 30 minutes following ingestion, 45 minutes following ingestion, 60 minutes following ingestion, and 90minutes following ingestion.
  Total ghrelin measured in blood via ELISA.

SECONDARY OUTCOMES:
Subjective appetite perception | Pre-ingestion, 30 minutes following ingestion, 45 minutes following ingestion, 60 minutes following ingestion, and 90minutes following ingestion.
  Measured using visual analogue scale
Free-living energy intake | Day 1 (day before the experimental session), Day 2 (day of the experimental session), and Day 3 (day after the experimental session).
  Free-living energy intake measured using a mobile application Keenoa

CONTACTS AND LOCATIONS:
Overall Officials: Tom J Hazell, PhD, Principal Investigator — Wilfrid Laurier University

IPD SHARING:
Plan to Share IPD: No